CLINICAL TRIAL: NCT02488915
Title: ARISE II (Analysis of Revascularization in Ischemic Stroke With EmboTrap) Study
Brief Title: Analysis of Revascularization in Ischemic Stroke With EmboTrap
Acronym: ARISEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuravi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP002
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Stroke; Ischemia
Keywords: Brain; Brain Clot; Brain Diseases; Brain Infarction; Cerebral Ischemia; Cerebrovascular Disorders; EmboTrap® Revascularization Device; EmboTrap; Ischemia; Ischemic; Ischemic Stroke; Mechanical Thrombectomy; Neurovascular Intervention; Revascularization; Stent Retriever; Stroke; Vascular Diseases; Neuravi
MeSH Terms: conditions — Stroke; Ischemia; Brain Diseases; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Ischemic Stroke; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EmboTrap® Revascularization Device (Experimental): Mechanical Thrombectomy with EmboTrap
  Interventions: Device: EmboTrap® Revascularization Device

INTERVENTIONS:
Device: EmboTrap® Revascularization Device
  Other Names: EmboTrap II

SUMMARY:
The study objective is to examine the recanalization efficacy of the EmboTrap device and its associated performance characteristics and to record associated clinical outcomes in a manner that facilitates relevant comparison of outputs with that of devices approved in the U.S. for clearing Large Vessel Occlusions.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or the patient's legally authorized representative has signed and dated an Informed Consent Form.
2. Aged between 18 years and 85 years (inclusive).
3. A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
4. NIHSS score ≥8 and ≤25.
5. Pre-ictal mRS score of 0 or 1.
6. The interventionalist estimates that at least one deployment of the EmboTrap device can be completed within 8 hours from the onset of symptoms.
7. Patients for whom IV-tPA is indicated and who are available for treatment, are treated with IV-tPA.
8. IV-tPA, if used, was initiated within 3 hrs of stroke onset (onset time is defined as the last time when the patient was witnessed to be at baseline), with investigator verification that the subject has received/is receiving the correct IV t-PA dose for the estimated weight.
9. Angiographic confirmation of an occlusion of an ICA (including T or L occlusions), M1 or M2 MCA, VA, or BA with mTICI flow of 0 - 1.
10. For strokes in the anterior circulation the following imaging criteria should also be met:

    1. MRI criterion: volume of diffusion restriction visually assessed ≤50 mL. OR
    2. CT criterion: ASPECTS 6 to 10 on baseline CT or CTA-source images, or, volume of significantly lowered CBV ≤50 mL.
11. The patient is indicated for neurothrombectomy treatment by the interventionalist and it is confirmed by diagnostic angiography that the device will be able to reach the target lesion proximally.

Exclusion Criteria:

1. Life expectancy likely less than 6 months.
2. Females who are pregnant or breastfeeding.
3. History of severe allergy to contrast medium.
4. Known nickel allergy at time of treatment.
5. Known current use of cocaine at time of treatment.
6. Patient has suffered a stroke in the past 3 months.
7. The patient presents with an NIHSS score <8 or >25 or is physician assessed as being in a clinically relevant uninterrupted coma.
8. Subject participating in another study involving an investigational device or drug.
9. Use of warfarin anticoagulation or any Novel Anticoagulant with International Normalized Ratio (INR) >3.0.
10. Platelet count <50,000/μL.
11. Glucose <50 mg/dL.
12. Any known hemorrhagic or coagulation deficiency.
13. Unstable renal failure with serum creatinine >3.0 or Glomerular Filtration Rate (GFR) <30.
14. Patients who have received a direct thrombin inhibitor within the last 48 hours; must have a partial thromboplastin time (PTT) less than 1.5 times the normal to be eligible.
15. All patients with severe hypertension on presentation (SBP> 220mmHg and/or DBP>120mmHg). All patients, in whom intravenous therapy with blood pressure medications is indicated, with hypertension that remains severe and sustained despite intravenous therapy (SBP >185mmHg and/or DBP>110mmHg). .
16. Known cerebral vasculitis.
17. Rapidly improving neurological status.
18. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
19. Ongoing seizure due to stroke.
20. Evidence of active systemic infection.
21. Known cancer with metastases.
22. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
23. Baseline computed tomography (CT) or MRI showing mass effect or intracranial tumor (except small meningioma).
24. Suspicion of aortic dissection, presumed septic embolus, or suspicion of bacterial endocarditis.
25. Stenosis, or any occlusion, in a proximal vessel that requires treatment or prevents access to the site of occlusion.
26. Evidence of dissection in the extra or intracranial cerebral arteries.
27. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Sam Zaidat, M.D., Principal Investigator — St. Vincent Mercy Mercy Hospital, Toledo,Ohio, USA; Prof. Tommy Andersson, M.D., Principal Investigator — Karolinska Institutet; Prof. Jeffery Saver, M.D., Study Director — UCLA, CA, USA.; Prof. Heinrich Mattle, M.D., Study Director — University of Berne, Berne, Switzerland.
Locations (12):
- United States (9):
  - UCLA, Los Angeles, California
  - Good Samaritan Hospital and Regional Medical Center, San Jose, California
  - University of Miami and Jackson Memorial Hospital, Miami, Florida
  - Emory University School of Medicine,, Atlanta, Georgia
  - Riverside Radiology and Interventional Associates, Columbus, Ohio
  - St Vincent Mercy Hospital, Toledo, Ohio
  - OHSU Stroke Center, Portland, Oregon
  - UPMC Stroke Center, Pittsburgh, Pennsylvania
  - Tennessee Interventional and Imaging Associates, Chattanooga, Tennessee
- AZ Groeninge, Kortrijk, Belgium
- UKSH Campus Kiel, Kiel, Germany
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo AJ, Soomro J, Andersson T, Saver JL, Ribo M, Bozorgchami H, Dabus G, Liebeskind DS, Jadhav A, Mattle H, Zaidat OO. Benchmarking the Extent and Speed of Reperfusion: First Pass TICI 2c-3 Is a Preferred Endovascular Reperfusion Endpoint. Front Neurol. 2021 May 11;12:669934. doi: 10.3389/fneur.2021.669934. eCollection 2021. PMID 34046008
- [Derived] Zaidat OO, Bozorgchami H, Ribo M, Saver JL, Mattle HP, Chapot R, Narata AP, Francois O, Jadhav AP, Grossberg JA, Riedel CH, Tomasello A, Clark WM, Nordmeyer H, Lin E, Nogueira RG, Yoo AJ, Jovin TG, Siddiqui AH, Bernard T, Claffey M, Andersson T. Primary Results of the Multicenter ARISE II Study (Analysis of Revascularization in Ischemic Stroke With EmboTrap). Stroke. 2018 May;49(5):1107-1115. doi: 10.1161/STROKEAHA.117.020125. Epub 2018 Apr 11. PMID 29643261

RESULTS

PARTICIPANT FLOW:
Groups:
- EmboTrap® Revascularization Device: Mechanical Thrombectomy with EmboTrap
  EmboTrap® Revascularization Device
Period: Overall Study
Arm/Group | EmboTrap® Revascularization Device
Started | 228
Completed | 202
Not Completed | 26
Not completed — Death | 21
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One subject enrolled was not treated with any thrombectomy device due to severe agitation.
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 206
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 17
  United States | 101
  Ireland | 6
  Germany | 43
  Spain | 35
  France | 23
  Switzerland | 2
National Institutes of Health Stroke Scale (NIHSS) Score [Mean (Standard Deviation); unit: Scores on a scale] — The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
  Scores on a scale | 15.8 (5)
Pre-stroke Modified Rankin Scale (mRS) [Count of Participants; unit: Participants] — mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. mRS scores range from 0 to 6:
  mRS 0 = No symptoms.
  mRS 1 = No significant disability.
  mRS 2 = Slight disability.
  mRS 3 = Moderate disability.
  mRS 4 = Moderately severe disability.
  mRS 5 = Severe disability.
  mRS 6 = Dead.
  Participants
    mRS 0 | 177
    mRS 1 | 49
    mRS 2 | 1
BMI [Mean (Standard Deviation); unit: kg per square meter] — Population: BMI not recorded per standard of care at all study sites
  kg per square meter
    number analyzed (Participants) | 166
    (all) | 28.7 (6)
Medical History [Count of Participants; unit: Participants]
  Previous Stroke/TIA | 43
  Previous MI/CAD | 45
  Atrial Fibrillation | 90
  Hypertension | 155
  Diabetes Mellitus | 45
  Dyslipidaemia | 98
  Current or ex-smoker | 56
Most Proximal occlusion location [Count of Participants; unit: Participants]
  Internal carotid artery | 10
  Internal carotid artery Terminus (L or T-type) | 25
  M1 middle cerebral artery | 126
  M2 middle cerebral artery | 57
  Other | 9

OUTCOME MEASURES:

1. Primary Outcome: Successful Revascularization Measured Using Modified Thrombolysis in Cerebrovascular Infarction (mTICI Inclusive of the 2c Rating)
Description: Successful achievement of the endpoint is defined as achieving an mTICI score of 2b or greater in the target vessel following 3 or less passes of the EmboTrap device. Patients treated with rescue prior to completion of three passes with EmboTrap were treated as failures to meet the primary revascularization endpoint. (Post measurement of the primary endpoint some patients subsequently received additional treatment.)
  -
  mTICI is a 6-point grading system for determining the response of thrombolytic therapy for ischaemic stroke:
  mTICI 0 = No perfusion
  mTICI 1 = Penetration but not perfusion
  mTICI 2a = Some perfusion with distal branch filling of <50% of territory visualized
  mTICI 2b = Substantial perfusion with distal branch filling of ≥50% of territory visualized
  mTICI 2c = Near-complete perfusion
  mTICI 3 = Complete perfusion
Time Frame: Post-treatment
Population: Analysis population includes all patients enrolled and treated with the EmboTrap device (N=227) irrespective of whether they met all incl/excl criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 182

2. Primary Outcome: Occurrence of Symptomatic Intracerebral Hemorrhage (sICH) Within 24 Hours Post-procedure and Any Other Serious Adverse Device Effects (SADE)
Description: The primary safety endpoint will be measured as the occurrence of Symptomatic Intracerebral hemorrhage (sICH) within 24 hours (-8/+12 hrs) post-procedure, together with any other Serious Adverse Device Effects (excluding those already counted in sICH).
  sICH was assessed using the Heidelberg Bleeding Classification, i.e. any intracerebral hemorrhage associated with an increase of ≥4 points in the NIHSS scale or an increase of ≥2 points of a NIHSS subcategory or that leads to major medical intervention. SADE was categorized as any serious adverse event that was deemed to be caused by the study device.
Time Frame: 24(-8/+12 hrs) hours post-procedure and 90(±14) days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 12

3. Secondary Outcome: Good Clinical Outcome as Defined by Modified Rankin Scale (mRS) Score ≤2
Description: Good Clinical Outcome is defined as achieving an mRS score of ≤2 at 90 days post procedure.
  -
  mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. mRS scores range from 0 to 6:
  mRS 0 = No symptoms.
  mRS 1 = No significant disability.
  mRS 2 = Slight disability.
  mRS 3 = Moderate disability.
  mRS 4 = Moderately severe disability.
  mRS 5 = Severe disability.
  mRS 6 = Dead.
Time Frame: 90(±14) days Post Procedure
Population: All patients enrolled and treated with the EmboTrap device for whom there is known data, including those who were subsequently treated with other therapies. However, outcome data excludes cases where the patient withdrew consent or was lost to follow up, with undefined/unknown scores.
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 217
Participants | 146

4. Secondary Outcome: Procedure Time
Description: The time from groin puncture to achievement of mTICI ≥2b, or if not obtained, to the final angiogram.
  -
  mTICI is a 6-point grading system for determining the response of thrombolytic therapy for ischaemic stroke:
  mTICI 0 = No perfusion
  mTICI 1 = Penetration but not perfusion
  mTICI 2a = Some perfusion with distal branch filling of <50% of territory visualized
  mTICI 2b = Substantial perfusion with distal branch filling of ≥50% of territory visualized
  mTICI 2c = Near-complete perfusion
  mTICI 3 = Complete perfusion
Time Frame: Post-treatment
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
minutes | 35 [24 to 58]

5. Secondary Outcome: All Procedure-related Mortality
Description: Any death that is deemed to have been caused by the study procedure.
Time Frame: Day 7 post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 0

6. Secondary Outcome: All-cause Mortality
Description: Any death that occurs within 90(±14) days post-procedure.
Time Frame: 90(±14) days Post Procedure
Population: Denominator excludes missing data. Participants who were Lost to Follow-up and Withdrew Consent were treated as missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 222
Participants | 20

7. Secondary Outcome: Occurrence of Serious Adverse Device Effects (SADE)
Description: SADE was categorized as any serious adverse event that was deemed to be caused by the study device.
Time Frame: 90(±14) days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 0

8. Secondary Outcome: Occurrence of Procedure Related Serious Adverse Events (PRSAE)
Description: PRSAE was categorized as any serious adverse event that was deemed to be caused by the study procedure.
Time Frame: 90(±14) days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 11

9. Secondary Outcome: Occurrence of Symptomatic Intracerebral Hemorrhage (sICH)
Description: sICH was assessed using the Heidelberg Bleeding Classification, i.e. any intracerebral hemorrhage associated with an increase of ≥4 points in the NIHSS scale or an increase of ≥2 points of a NIHSS subcategory or that leads to major medical intervention.
Time Frame: 24(-8/+12) hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 12

10. Secondary Outcome: Occurrence of Neurological Deterioration
Description: An increase of 4 points or more on the National Institutes of Health Stroke Scale (NIHSS) at 24 hours (-8/+12 hrs) post-procedure. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
Time Frame: 24(-8/+12) hours post-procedure
Population: Denominator exclude missing data. Participant who were not assessed for NIHSS at 24hrs and/or those who used rescue therapy at any time during the procedure were treated as missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 178
Participants | 8

11. Secondary Outcome: Proportion of Subjects With Evidence of Infarction of a Previously Uninvolved Vascular Territory
Description: Infarction (i.e. brain tissue death) of a previously uninvolved vascular territory (i.e. region of the brain) is evaluated from 24-hour imaging (Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)).
Time Frame: 24(-8/+12) hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 34

12. Secondary Outcome: Time to Treat
Description: The time from first baseline angiogram to achievement of mTICI ≥2b, or if not obtained, to the final angiogram.
  -
  mTICI is a 6-point grading system for determining the response of thrombolytic therapy for ischaemic stroke:
  mTICI 0 = No perfusion
  mTICI 1 = Penetration but not perfusion
  mTICI 2a = Some perfusion with distal branch filling of <50% of territory visualized
  mTICI 2b = Substantial perfusion with distal branch filling of ≥50% of territory visualized
  mTICI 2c = Near-complete perfusion
  mTICI 3 = Complete perfusion
Time Frame: Post-treatment
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
minutes | 24 [13 to 45]

13. Post Hoc Outcome: Proportion of Subjects With New Territory Embolisation
Description: Embolisation of any new territories was recorded directly post-treatment.
Time Frame: Post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 227
Participants | 15

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | EmboTrap® Revascularization Device
All-Cause Mortality (participants affected / at risk) | 20/227
Serious Adverse Events (participants affected / at risk) | 92/227
Other Adverse Events (participants affected / at risk) | 175/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EmboTrap® Revascularization Device (N=227)
Myocardial infarction (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Vessel puncture site thrombosis (General disorders) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Septic shock (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 15 (15)
Ischaemic stroke (Nervous system disorders) | 14 (14)
Brain oedema (Nervous system disorders) | 7 (7)
Neurological decompensation (Nervous system disorders) | 5 (5)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4)
Seizure (Nervous system disorders) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 3 (3)
Carotid artery dissection (Nervous system disorders) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 2 (2)
Vessel perforation (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EmboTrap® Revascularization Device (N=227)
Atrial fibrillation (Cardiac disorders) | 17 (18)
Urinary tract infection (Infections and infestations) | 30 (30)
Haemorrhagic transformation stroke (Nervous system disorders) | 54 (55)
Subarachnoid haemorrhage (Nervous system disorders) | 28 (28)
Headache (Nervous system disorders) | 19 (19)
Cerebral vasoconstriction (Nervous system disorders) | 12 (12)
Hypotension (Vascular disorders) | 14 (14)
Hypertension (Vascular disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02488915/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02488915/SAP_001.pdf